CLINICAL TRIAL: NCT00763893
Title: Multicenter, Randomised, Double Blind Study of the Efficacy of Losartan on Aortic Dilatation in Patients With Marfan Syndrome
Brief Title: Study of the Efficacy of Losartan on Aortic Dilatation in Patients With Marfan Syndrome
Acronym: MARFANSARTAN
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: A similar publication has been released, suggesting a beneficial effect of sartans, and only 15 patients remained to be seen for their visit at 36 months.
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: P060210; 2006-006112-30 (EudraCT Number)
Record Dates: First submitted 2008-09-30; First posted 2008-10-01 (Estimated); Last update posted 2015-11-04 (Estimated); Status verified 2015-10

CONDITIONS: Marfan Syndrome
Keywords: Marfan syndrome; Angiotensin II Type 1 Receptor Blockers; Aortic Aneurysm, Thoracic
MeSH Terms: conditions — Marfan Syndrome; Aortic Aneurysm, Thoracic | interventions — Losartan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A: Placebo (Placebo Comparator): placebo
  Interventions: Drug: placebo
- B: Losartan (Active Comparator): Losartan
  Interventions: Drug: Losartan

INTERVENTIONS:
Drug: placebo — Cover key details of the intervention. Must be sufficiently detailed to distinguish between arms of a study (e.g., comparison of different dosages of drug) and/or among similar interventions (e.g., comparison of multiple implantable cardiac defibrillators). For example, interventions involving drugs may include dosage form, dosage, frequency and duration.
  Arms: A: Placebo
Drug: Losartan — 50 mg/day if < weight 50 kg 100 mg/day if weight > 50 kg
  Arms: B: Losartan

SUMMARY:
The purpose of this study is to evaluate if losartan limits aortic dilatation in patients with Marfan syndrome.

DETAILED DESCRIPTION:
Aim : evaluate the efficacy of losartan for limiting aortic dilatation in patients with marfan syndrome receiving standard therapy

Inclusion criteria :

10 years or older Marfan syndrome according to international criteria Signed informed consent

Non inclusion :

Previous surgery of the ascending aorta, or surgery planned Non echogenicity Contre-indication lactose Pregnancy on going or planned within 3 years Breast feeding Participation in another clinical study Non member of the social security or CMU

Number of subjects : the number of subjects (150 per group) is derived from the study from Shores et al (1994) demonstrating the benefit of beta-blockade in Marfan patient and uses a decrease by half of the aortic dilatation with losartan

Follow-up is 3 years, after inclusion period of 2 years. A total of 5 years is expected

Methods : randomised double blind vs placebo study. All French centres de competence for marfan syndrome and the centre de reference are participating in the study.

End points : main endpoint is evolution of normalised aortic diameter. Secondary endpoints include clinical events (cardiac surgery or aortic dissection, hospitalisation in cardiology department, death), tolerance of the drug, and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* 10 years or older
* Marfan syndrome according to international criteria Signed informed consent

Exclusion Criteria:

* Previous surgery of the ascending aorta, or surgery planned
* Non echogenicity
* Contre-indication lactose
* Pregnancy on going or planned within 3 years
* Breast feeding
* Participation in another clinical study
* Non member of the social security or CMU

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 303 (Actual)
Dates: Start 2008-09; Primary Completion 2014-01 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
normalised aortic diameter at the level of the sinus of valsalva | every six months

SECONDARY OUTCOMES:
cardiac surgery, hospitalisation in cardiology ward, death | during the follow up

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume JONDEAU, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Bichat, Paris, France

REFERENCES:
- [Result] Detaint D, Aegerter P, Tubach F, Hoffman I, Plauchu H, Dulac Y, Faivre LO, Delrue MA, Collignon P, Odent S, Tchitchinadze M, Bouffard C, Arnoult F, Gautier M, Boileau C, Jondeau G. Rationale and design of a randomized clinical trial (Marfan Sartan) of angiotensin II receptor blocker therapy versus placebo in individuals with Marfan syndrome. Arch Cardiovasc Dis. 2010 May;103(5):317-25. doi: 10.1016/j.acvd.2010.04.008. Epub 2010 Jul 1. PMID 20619242
- [Result] Milleron O, Arnoult F, Ropers J, Aegerter P, Detaint D, Delorme G, Attias D, Tubach F, Dupuis-Girod S, Plauchu H, Barthelet M, Sassolas F, Pangaud N, Naudion S, Thomas-Chabaneix J, Dulac Y, Edouard T, Wolf JE, Faivre L, Odent S, Basquin A, Habib G, Collignon P, Boileau C, Jondeau G. Marfan Sartan: a randomized, double-blind, placebo-controlled trial. Eur Heart J. 2015 Aug 21;36(32):2160-6. doi: 10.1093/eurheartj/ehv151. Epub 2015 May 2. PMID 25935877
- [Derived] Jiang P, Loyau S, Tchitchinadze M, Ropers J, Jondeau G, Jandrot-Perrus M. Inhibition of Glycoprotein VI Clustering by Collagen as a Mechanism of Inhibiting Collagen-Induced Platelet Responses: The Example of Losartan. PLoS One. 2015 Jun 8;10(6):e0128744. doi: 10.1371/journal.pone.0128744. eCollection 2015. PMID 26052700